CLINICAL TRIAL: NCT05087992
Title: A Phase Ia/Ib, Open Label, Multicentre, Dose Escalation Study of BI 905711 in Combination With Chemotherapy Followed by Expansion Cohorts in Patients With Advanced Gastrointestinal Cancers
Brief Title: A Study to Find the Best Dose of BI 905711 in Combination With Chemotherapy and to Test Whether This Dose Helps People With Advanced Gastrointestinal Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1412-0003; 2021-003041-37 (EudraCT Number)
Record Dates: First submitted 2021-10-11; First posted 2021-10-21 (Actual); Results first posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Gastrointestinal Cancer, Metastatic
MeSH Terms: conditions — Gastrointestinal Neoplasms; Neoplasm Metastasis | interventions — IFL protocol; Bevacizumab

STUDY DESIGN:
Intervention Model Description: Phase 1a non randomized, Phase 1b randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 0.6 mg/kg BI 905711 + FOLFIRI + bevacizumab (Experimental): Patients with colorectal adenocarcinoma (CRC) received a single administration of 0.6 milligrams (mg) / kilograms (kg) of BI 905711 intravenously on Day 3 of each 14-day cycle. Patients also received FOLFIRI (irinotecan: 180 mg/squaremeters (m2) over 1.5 hours (hrs), leucovorin: 400 mg/m2 (in Japan: levoleucovorin: 200 mg/m2) over 2 hrs, fluorouracil: 400 mg/m2 bolus or 2400 mg/m2 46 hrs continuous infusion) in combination with bevacizumab, 5 mg/kg over 30 minutes (min) intravenously on Day 1 of each 14-day cycle.
  Interventions: Drug: BI 905711; Drug: FOLFIRI; Drug: Bevacizumab
- 1.2 mg/kg BI 905711 + FOLFIRI + bevacizumab (Experimental): Patients with colorectal adenocarcinoma (CRC) received a single administration of 1.2 mg/kg of BI 905711 intravenously on Day 3 of each 14-day cycle. Patients also received FOLFIRI (irinotecan: 180 mg/m2 over 1.5 hours (hrs), leucovorin: 400 mg/m2 (in Japan: levoleucovorin: 200 mg/m2) over 2 hrs, fluorouracil: 400 mg/m2 bolus or 2400 mg/m2 46 hrs continuous infusion) in combination with bevacizumab, 5 mg/kg over 30 minutes (min) intravenously on Day 1 of each 14-day cycle.
  Interventions: Drug: BI 905711; Drug: FOLFIRI; Drug: Bevacizumab
- FOLFIRI + bevacizumab (Active Comparator): Patients with colorectal adenocarcinoma (CRC) received FOLFIRI (irinotecan: 180 mg/m2 over 1.5 hours (hrs), leucovorin [or levoleucovorin]: 400 mg/m2 (in Japan: levoleucovorin: 200 mg/m2) over 2 hrs, fluorouracil: 400 mg/m2 bolus or 2400 mg/m2 46 hrs continuous infusion) in combination with bevacizumab, 5 mg/kg over 30 minutes (min) intravenously on Day 1 of each 14-day cycle.
  Interventions: Drug: FOLFIRI; Drug: Bevacizumab

INTERVENTIONS:
Drug: BI 905711 — BI 905711
  Arms: 0.6 mg/kg BI 905711 + FOLFIRI + bevacizumab; 1.2 mg/kg BI 905711 + FOLFIRI + bevacizumab
Drug: FOLFIRI — FOLFIRI
Drug: Bevacizumab — Bevacizumab

SUMMARY:
This study is open to adults with advanced colorectal cancer or with advanced pancreatic cancer. The study has 2 parts. In the first part, participants with colorectal cancer get a medicine called BI 905711 combined with chemotherapy and bevacizumab. The purpose of the first part is to find the highest BI 905711 dose participants can tolerate. In the second part, participants with colorectal cancer or pancreatic cancer get BI 905711 combined with chemotherapy. Some participants also get bevacizumab. The second part tests whether BI 905711 makes tumours shrink. Participants get BI 905711, chemotherapy and bevacizumab about every 2 weeks as an infusion into a vein. Participants can stay in the study as long as they benefit from treatment and can tolerate it. The doctors regularly check the health of the participants and note any health problems that could have been caused by the study treatment. The doctors also monitor the size of the tumour.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent in accordance with International Council of Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial.
* Of legal adult age (according to local legislation) at screening.
* Histologically or cytologically confirmed, advanced unresectable or metastatic colorectal adenocarcinoma.
* Colorectal adenocarcinoma (CRC): Patients who have Progressive disease (PD) after prior oxaliplatin-based first line therapy or within 6 months after the end of oxaliplatin-based adjuvant therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1.
* Life expectancy ≥ 3 months in the opinion of the investigator.
* Availability and willingness to provide tumor tissue (fresh biopsy or archival) for biomarker analysis. Only non-significant risk procedures per the investigator's judgment will be used to obtain any biopsies specified in this study. In case a fresh tumor biopsy cannot be obtained, the recruitment of the patient may proceed on a case-by-case basis after agreement between the investigator and BI. In such a case, an archived tumor tissue specimen must be submitted.
* Adequate hepatic, pancreatic, renal and bone marrow functions as defined by all of the below:

  * Total bilirubin ≤ 1.5 x institutional upper level of normal (ULN).
  * Alanine transaminase (ALT) and Aspartate transaminase (AST) ≤2.5 x institutional ULN or ≤5 x institutional ULN for patients with known liver metastases.
  * Serum creatinine ≤1.5x institutional ULN. If creatinine is > 1.5 x ULN, patient is eligible if concurrent creatinine clearance ≥ 50 ml/min (≥ 0.05L/min) (measured or calculated by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula or Japanese version of CKD-EPI formula for Japanese patients).
  * Absolute neutrophil count (ANC) ≥ 1.5 x 1^9/L, ≥ 1.5 x 10^3/μL, or ≥ 1500/mm^3
  * Platelets ≥ 100 x 10^9/L, ≥ 100 x 10^3/μL, or ≥ 100 x 10^3/mm^3
  * Hemoglobin (Hb) ≥ 8.5 g/dl, ≥ 85 g/L, or ≥ 5.3 mmol/L (without transfusion within previous week) Serum lipase ≤ 1.5 institutional ULN (Only for CRC cohort); >1.5 - 2.0 x ULN or asymptomatic >2.0 - 5.0 x ULN if related to Pancreatic Ductal Adenocarcinoma (PDAC) (Only for PDAC cohort) Further inclusion criteria apply.

Exclusion criteria:

* Any prior irinotecan-based therapy in the metastatic setting.
* Previous systemic anti-cancer therapy within the specified timeframe from the last dose intake to the first dose of trial treatment as follows:

  * Any non-investigational drug, including anti-angiogenic agents (bevacizumab or ramucirumab or aflibercept) and anti-EGFR antibodies (cetuximab or panitumumab), within 14 days.
  * Any investigational drug or other antibodies including immune checkpoint inhibitors, within 28 days.
* Currently enrolled in another investigational device or drug trial. Patients who are in follow-up/observation for another clinical trial are eligible.
* Radiation therapy within 4 weeks prior to start of treatment. However, palliative radiotherapy for symptomatic metastasis is allowed if completed within 2 weeks prior to start of treatment.
* Any serious concomitant disease or medical condition affecting compliance with trial requirements or which are considered relevant for the evaluation of the efficacy or safety of the trial drug, such as neurologic, psychiatric, infectious disease or active ulcers (gastro-intestinal (GI) tract, skin) or laboratory abnormality that may increase the risk associated with trial participation or trial drug administration, and in the judgment of the Investigator, would make the patient inappropriate for entry into the trial.
* Known pathological condition of GI tract, liver and pancreas, excluding the disease under study, that may interfere with assessment of drug safety or may increase the risk of toxicity:

  * inflammatory bowel disease
  * chronic pancreatitis
  * other serious GI pathological conditions by judgment of the investigator e.g. autoimmune disease with GI involvement, unexplained active diarrhea CTCAE v5.0 grade ≥ 2.
* Known history of human immunodeficiency virus (HIV) infection.
* Any of the following laboratory evidence of hepatitis virus infection. Test results obtained in routine diagnostics are acceptable if done within 14 days before the informed consent date:

  * Positive results of hepatitis B surface (HBs) antigen
  * Presence of HBc antibody together with hepatitis B virus deoxyribonucleic acid (HBV-DNA)
  * Presence of hepatitis C ribonucleic acid (RNA) Further exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-11-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States
- UZ Leuven, Leuven, Belgium
- Beijing Cancer Hospital, Beijing, China
- HOP la Milétrie, Poitiers, France
- National Cancer Center Hospital East, Chiba, Kashiwa, Japan

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The main objective of this phase Ia/Ib, open label, multicentre, dose escalation followed by expansion cohorts study was to determine the maximum tolerated dose (MTD) and the recommended dose for expansion (RDE), and to explore the pharmacokinetics, pharmacodynamics, safety and efficacy of BI 905711 in combination with FOLFIRI regimen plus bevacizumab in colorectal adenocarcinoma (CRC) patients.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | 0.6 mg/kg BI 905711 + FOLFIRI + Bevacizumab | 1.2 mg/kg BI 905711 + FOLFIRI + Bevacizumab | FOLFIRI + Bevacizumab
Started | 9 | 3 | 1
Completed | 0 | 0 | 1
Not Completed | 9 | 3 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — clinical disease progression | 3 | 1 | 0
Not completed — objective disease progression | 4 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This included all subjects who were dispensed study medication and were documented to have been treated with at least one dose of BI 905711 or chemotherapy. This TS was used for both safety and efficacy analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.6 mg/kg BI 905711 + FOLFIRI + Bevacizumab | 1.2 mg/kg BI 905711 + FOLFIRI + Bevacizumab | FOLFIRI + Bevacizumab | Total
Number analyzed (Participants) | 9 | 3 | 1 | 13
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.4 (10.7) | 60.3 (11.2) | NA — data protection, only 1 patient | 54.6 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | NA — data protection, only 1 patient | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | 4 | 2 | NA — data protection, only 1 patient | NA — Total not calculated because data are not available (NA) in one or more arms.
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | NA — data protection, only 1 patient | NA — Total not calculated because data are not available (NA) in one or more arms.
  Not Hispanic or Latino | 9 | 3 | NA — data protection, only 1 patient | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 0 | 0 | NA — data protection, only 1 patient | NA — Total not calculated because data are not available (NA) in one or more arms.
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | NA — data protection, only 1 patient | NA — Total not calculated because data are not available (NA) in one or more arms.
  Asian | 5 | 1 | NA — data protection, only 1 patient | NA — Total not calculated because data are not available (NA) in one or more arms.
  Native Hawaiian or Other Pacific Islander | 0 | 2 | NA — data protection, only 1 patient | NA — Total not calculated because data are not available (NA) in one or more arms.
  Black or African American | 0 | 0 | NA — data protection, only 1 patient | NA — Total not calculated because data are not available (NA) in one or more arms.
  White | 4 | 0 | NA — data protection, only 1 patient | NA — Total not calculated because data are not available (NA) in one or more arms.
  More than one race | 0 | 0 | NA — data protection, only 1 patient | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 0 | 0 | NA — data protection, only 1 patient | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Determination of the Maximum Tolerated Dose (MTD) of BI 905711
Description: Maximum tolerated dose (MTD) was defined as the highest dose with less than 25% risk of the true dose-limiting toxicity (DLT) rate being equal or above 33% during the MTD evaluation period.
  The MTD was to be considered reached if one of the following criteria was fulfilled: the posterior probability of the true DLT rate in the target interval (0.16, 0.33) of the MTD was above 0.5, or at least 12 patients had been treated in Phase Ia, of which at least 6 at the MTD.
Time Frame: From cycle 1 Day 1 until the day before cycle 3 Day 1 (2 14-day treatment cycles), or end of the residual effect period (REP) (30 days + 5 days) in case of discontinuation before start of cycle 3, up to 35 days.
Population: Maximum tolerated dose evaluation set (MTDS): This included all patients in the TS who were not replaced for the MTD determination. The MTDS was used for the primary analyses of dose-limiting toxicities (DLTs) and MTD determination.
Measure: Number; unit: milligram / kilogram (mg/kg)
Groups:
- BI 905711 + FOLFIRI + Bevacizumab: Comprises all dose cohorts during the dose escalation phase. Patients with colorectal adenocarcinoma (CRC) received a single administration of 0.6 or 1.2 mg/kg of BI 905711 intravenously on Day 3 of each 14-day cycle. Patients also received FOLFIRI (irinotecan: 180 mg/m2 over 1.5 hours (hrs), leucovorin [or levoleucovorin]: 400 mg/m2 (in Japan: levoleucovorin: 200 mg/m2) over 2 hrs, fluorouracil: 400 mg/m2 bolus or 2400 mg/m2 46 hrs continuous infusion) in combination with bevacizumab, 5 mg/kg over 30 minutes (min) intravenously on Day 1 of each 14-day cycle.
Arm/Group | BI 905711 + FOLFIRI + Bevacizumab
Number analyzed (Participants) | 12
milligram / kilogram (mg/kg) | NA — Criteria for reaching MTD were not fulfilled.

2. Primary Outcome: Number of Patients With Dose Limiting Toxicity (DLT) During MTD Evaluation
Description: Number of patients with dose limiting toxicity (DLT) during MTD evaluation is presented.
Time Frame: From cycle 1 Day 1 until the day before cycle 3 Day 1 (2 14-day treatment cycles), or end of the REP (30 days + 5 days) in case of discontinuation before start of cycle 3, up to 35 days.
Population: Maximum tolerated dose evaluation set (MTDS): This included all patients in the TS who were not replaced for the MTD determination. The MTDS was used for the primary analyses of dose-limiting toxicities (DLTs) and MTD determination. Only treated patients from the dose escalation part were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.6 mg/kg BI 905711 + FOLFIRI + Bevacizumab | 1.2 mg/kg BI 905711 + FOLFIRI + Bevacizumab
Number analyzed (Participants) | 6 | 3
Participants | 0 | 2

3. Primary Outcome: Confirmed Objective Response (OR)
Description: Confirmed objective response (OR) as assessed by the investigator based on Response Evaluation Criteria in Solid Tumors (RECIST 1.1) for target lesions and assessed by MRI in patients with measurable disease, defined as the best overall response of complete response (CR) or partial response (PR), from the first administration of trial medication until the earliest of progressive disease (PD), death or last evaluable tumor assessment before start of subsequent anti-cancer therapy.
Time Frame: From the first administration of trial medication until the earliest of progressive disease (PD), death or last evaluable tumor assessment before start of subsequent anti-cancer therapy, up to 54 weeks.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | 0.6 mg/kg BI 905711 + FOLFIRI + Bevacizumab | 1.2 mg/kg BI 905711 + FOLFIRI + Bevacizumab | FOLFIRI + Bevacizumab
Number analyzed (Participants) | 9 | 3 | 1
Participants | 0 | 0 | 0

4. Primary Outcome: Number of PDAC Patients With DLTs During the MTD Evaluation Period Assessed in the First 6 Patients
Description: In safety run-in part of Pancreatic Ductal Adenocarcinoma (PDAC) cohort. Number of PDAC patients with DLTs during the MTD evaluation period assessed in the first 6 patients is presented.
Time Frame: as for outcome 2
Population: Due to the stopping criteria in the protocol of the clinical development of BI 905711, recruitment in this trial was prematurely discontinued during the Phase Ib expansion phase and no PDAC patients were enrolled.
Groups:
- 0.6 mg/kg BI 905711 + FOLFIRI in Pancreatic Ductal Adenocarcinoma (PDAC) Expansion Cohort (Phase Ib): Patients with pancreatic ductal adenocarcinoma (PDAC) received a single administration of 0.6 mg/kg of BI 905711 intravenously on Day 3 of each 14-day cycle. Patients also received FOLFIRI (irinotecan: 70 or 180 mg/m2 over 1.5 hours (hrs), leucovorin [or levoleucovorin]: 400 mg/m2 (in Japan: levoleucovorin: 200 mg/m2) over 2 hrs, fluorouracil: 400 mg/m2 bolus or 2400 mg/m2 46 hrs continuous infusion) intravenously on Day 1 of each 14-day cycle.
Arm/Group | 0.6 mg/kg BI 905711 + FOLFIRI in Pancreatic Ductal Adenocarcinoma (PDAC) Expansion Cohort (Phase Ib)
Number analyzed (Participants) | 0

5. Secondary Outcome: Maximum Measured Plasma Concentration of BI 905711 During the First Cycle (Cmax)
Description: Maximum measured plasma concentration of BI 905711 during the first cycle (Cmax) in phase Ia is presented.
Time Frame: At 5 minutes (min) before start of BI 905711 infusion and at 30 min, 7 hours (hrs), 24 hrs, 48 hrs, 168 hrs and 336 hrs after BI 905711 infusion in cycle 1.
Population: Pharmacokinetic parameter analysis set (PKS): This included all subjects in the treated set (TS) who provided at least one PK endpoint and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms / milliliter (ng/ml)
Arm/Group | 0.6 mg/kg BI 905711 + FOLFIRI + Bevacizumab | 1.2 mg/kg BI 905711 + FOLFIRI + Bevacizumab
Number analyzed (Participants) | 9 | 3
nanograms / milliliter (ng/ml) | 6100 (36.6) | 11500 (23.9)

6. Secondary Outcome: Maximum Measured Plasma Concentration of BI 905711 After Multiple Cycles (Cmax)
Description: Maximum measured plasma concentration of BI 905711 after multiple cycles (Cmax) in phase Ia is presented.
Time Frame: Cycle 3: At 5 minutes (min) before start of BI 905711 infusion and at 30 min, 7 hours (hrs), 24 hrs, 48 hrs, 168 hrs and 336 hrs after BI 905711 infusion.
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/ml)
Arm/Group | 0.6 mg/kg BI 905711 + FOLFIRI + Bevacizumab | 1.2 mg/kg BI 905711 + FOLFIRI + Bevacizumab
Number analyzed (Participants) | 9 | 3
nanograms/milliliter (ng/ml) | 6660 (25.4) | 9280 (23.8)

7. Secondary Outcome: Area Under the Concentration-time Curve in Plasma of BI 905711 During the First Cycle (AUC0-336)
Description: Area under the concentration-time curve in plasma of BI 905711 during the first cycle (AUC0-336) in phase Ia is presented.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours * nanograms/milliliter (h*ng/ml)
Arm/Group | 0.6 mg/kg BI 905711 + FOLFIRI + Bevacizumab | 1.2 mg/kg BI 905711 + FOLFIRI + Bevacizumab
Number analyzed (Participants) | 8 | 3
hours * nanograms/milliliter (h*ng/ml) | 372000 (53.4) | 702000 (49.4)

8. Secondary Outcome: Area Under the Concentration Time-curve in Plasma of BI 905711 After Multiple Cycles (AUC0-336)
Description: Area under the concentration time-curve in plasma of BI 905711 after multiple cycles (AUC0-336) in phase Ia is presented.
Time Frame: as for outcome 6
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours * nanograms/milliliter (h*ng/ml)
Arm/Group | 0.6 mg/kg BI 905711 + FOLFIRI + Bevacizumab | 1.2 mg/kg BI 905711 + FOLFIRI + Bevacizumab
Number analyzed (Participants) | 8 | 3
hours * nanograms/milliliter (h*ng/ml) | 352000 (73.3) | 565000 (29.0)

9. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-Free Survival (PFS) defined from date of start of treatment to the date of disease progression or death, whichever is earlier as assessed by the investigator according to RECIST 1.1 is presented.
Time Frame: From date of start of treatment to the date of disease progression or death, whichever is earlier as assessed by the investigator according to RECIST 1.1., up to 54 weeks.
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | 0.6 mg/kg BI 905711 + FOLFIRI + Bevacizumab | 1.2 mg/kg BI 905711 + FOLFIRI + Bevacizumab | FOLFIRI + Bevacizumab
Number analyzed (Participants) | 9 | 3 | 1
weeks | 31.00 [8.43 to 39.29] | 29.57 [11.71 to 33.43] | NA [NA to NA] — Patient did not progress

10. Secondary Outcome: Maximum Percentage Change From Baseline in the Sum of Longest Target Lesion Diameters
Description: Radiological (CT Scan) tumor shrinkage, defined as the difference between the minimum post-baseline sum of longest diameters of target lesions and the baseline sum of longest diameters of the same set of target lesions according to RECIST 1.1. is presented.
  Negative values indicate a reduction in the sum of target lesion diameters and positive values indicate an increase. Median change from baseline was calculated for each patient and then summarized over all patients.
Time Frame: At baseline and every 8 weeks (± 7 days) until progression or start of further treatment for disease, up to 54 weeks.
Population: Treated set (TS): This included all subjects who were dispensed study medication and were documented to have been treated with at least one dose of BI 905711 or chemotherapy. This TS was used for both safety and efficacy analyses. Only patients with tumor diameter measurements were included.
Measure: Median (Inter-Quartile Range); unit: Percentage change in tumor diameter
Arm/Group | 0.6 mg/kg BI 905711 + FOLFIRI + Bevacizumab | 1.2 mg/kg BI 905711 + FOLFIRI + Bevacizumab | FOLFIRI + Bevacizumab
Number analyzed (Participants) | 8 | 3 | 0
Percentage change in tumor diameter | -13.9 [-28.3 to 18.6] | 4.5 [-21.7 to 6.3] |

11. Secondary Outcome: Duration of Objective Response (OR)
Description: The duration of OR is measured from the time measurement criteria are first met for complete response (CR)/ partial response (PR) (whichever is first recorded) until the first date that recurrent or progressive disease (PD) is objectively documented (taking as reference for PD the smallest measurements recorded on study) according to RECIST 1.1. .
Time Frame: From the time measurement criteria are first met for CR/PR (whichever is first recorded) until the first date that recurrent or PD is objectively documented, up to 54 weeks.
Population: Treated set (TS): This included all subjects who were dispensed study medication and were documented to have been treated with at least one dose of BI 905711 or chemotherapy. This TS was used for both safety and efficacy analyses. Only patients with objective response were included.
Arm/Group | 0.6 mg/kg BI 905711 + FOLFIRI + Bevacizumab | 1.2 mg/kg BI 905711 + FOLFIRI + Bevacizumab | FOLFIRI + Bevacizumab
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Disease Control
Description: Disease control, defined as complete response (CR), partial response (PR), or stable disease (SD) lasting at least 16 weeks according to RECIST 1.1 from the start of treatment until the earliest of PD, death or last evaluable tumor assessment and before start of subsequent anti-cancer therapy.
Time Frame: From the start of treatment until the earliest of PD, death or last evaluable tumor assessment and before start of subsequent anti-cancer therapy, up to 54 weeks.
Population: Treated set (TS): This included all subjects who were dispensed study medication and were documented to have been treated with at least one dose of BI 905711 or chemotherapy. This TS was used for both safety and efficacy analyses. Only patients with disease control were included.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | 0.6 mg/kg BI 905711 + FOLFIRI + Bevacizumab | 1.2 mg/kg BI 905711 + FOLFIRI + Bevacizumab | FOLFIRI + Bevacizumab
Number analyzed (Participants) | 6 | 2 | 0
days | 248.0 [120 to 325] | 220.5 [207 to 234] |

13. Secondary Outcome: Maximum Measured Plasma Concentration of BI 905711 During the First Cycle (Cmax) in Phase Ib
Description: Maximum measured plasma concentration of BI 905711 during the first cycle (Cmax) in phase Ib is presented.
Time Frame: as for outcome 5
Population: Due to the termination of the clinical development of BI 905711, recruitment in this trial was prematurely discontinued during the Phase Ib expansion phase and no PDAC patients were enrolled.
Arm/Group | 0.6 mg/kg BI 905711 + FOLFIRI + Bevacizumab | 1.2 mg/kg BI 905711 + FOLFIRI + Bevacizumab | 0.6 mg/kg BI 905711 + FOLFIRI in Pancreatic Ductal Adenocarcinoma (PDAC) Expansion Cohort (Phase Ib)
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Maximum Measured Plasma Concentration of BI 905711 After Multiple Cycles (Cmax) in Phase Ib
Description: Maximum measured plasma concentration of BI 905711 after multiple cycles (Cmax) in phase Ib is presented.
Time Frame: as for outcome 6
Population: as for outcome 13
Groups:
- 0.6 mg/kg BI 905711 + FOLFIRI in Pancreatic Ductal Adenocarcinoma (PDAC) Expansion Cohort: Patients with pancreatic ductal adenocarcinoma (PDAC) received a single administration of 0.6 mg/kg of BI 905711 intravenously on Day 3 of each 14-day cycle. Patients also received FOLFIRI (irinotecan: 70 or 180 mg/m2 over 1.5 hours (hrs), leucovorin [or levoleucovorin]: 400 mg/m2 (in Japan: levoleucovorin: 200 mg/m2) over 2 hrs, fluorouracil: 400 mg/m2 bolus or 2400 mg/m2 46 hrs continuous infusion) intravenously on Day 1 of each 14-day cycle.
Arm/Group | 0.6 mg/kg BI 905711 + FOLFIRI + Bevacizumab | 1.2 mg/kg BI 905711 + FOLFIRI + Bevacizumab | 0.6 mg/kg BI 905711 + FOLFIRI in Pancreatic Ductal Adenocarcinoma (PDAC) Expansion Cohort
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Area Under the Concentration-time Curve of BI 9057 During the First Treatment Cycle (AUC0-t2) in Phase Ib
Description: Area under the concentration-time curve of BI 9057 during the first treatment cycle (AUC0-t2) in phase Ib is presented.
Time Frame: as for outcome 5
Population: as for outcome 13
Arm/Group | 0.6 mg/kg BI 905711 + FOLFIRI + Bevacizumab | 1.2 mg/kg BI 905711 + FOLFIRI + Bevacizumab | 0.6 mg/kg BI 905711 + FOLFIRI in Pancreatic Ductal Adenocarcinoma (PDAC) Expansion Cohort (Phase Ib)
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Area Under the Concentration-time Curve of BI 9057 After Multiple Cycles (AUC0-t2) in Phase Ib
Description: Area under the concentration-time curve of BI 9057 after multiple cycles (AUC0-t2) in phase Ib is presented.
Time Frame: as for outcome 6
Population: as for outcome 13
Arm/Group | 0.6 mg/kg BI 905711 + FOLFIRI + Bevacizumab | 1.2 mg/kg BI 905711 + FOLFIRI + Bevacizumab | 0.6 mg/kg BI 905711 + FOLFIRI in Pancreatic Ductal Adenocarcinoma (PDAC) Expansion Cohort (Phase Ib)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 54 weeks.
Description: Treated set (TS): This includes all subjects who were dispensed study medication and were documented to have been treated with at least one dose of BI 905711 or chemotherapy. This TS is used for both safety and efficacy analyses.
Arm/Group | 0.6 mg/kg BI 905711 + FOLFIRI + Bevacizumab | 1.2 mg/kg BI 905711 + FOLFIRI + Bevacizumab | FOLFIRI + Bevacizumab
All-Cause Mortality (participants affected / at risk) | 3/9 | 2/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 4/9 | 2/3 | 0/1
Other Adverse Events (participants affected / at risk) | 9/9 | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.6 mg/kg BI 905711 + FOLFIRI + Bevacizumab (N=9) | 1.2 mg/kg BI 905711 + FOLFIRI + Bevacizumab (N=3) | FOLFIRI + Bevacizumab (N=1)
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0
Gastroenteritis Escherichia coli (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0
Oesophageal infection (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.6 mg/kg BI 905711 + FOLFIRI + Bevacizumab (N=9) | 1.2 mg/kg BI 905711 + FOLFIRI + Bevacizumab (N=3) | FOLFIRI + Bevacizumab (N=1)
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 5 | 3 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0
Catheter site inflammation (General disorders) | 1 | 0 | 0
Device related thrombosis (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 1
Influenza like illness (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 1 | 0
Pain (General disorders) | 2 | 0 | 0
Pyrexia (General disorders) | 3 | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1 | 0
Coronavirus infection (Infections and infestations) | 1 | 0 | 0
Rash pustular (Infections and infestations) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0
Tongue fungal infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Stoma site inflammation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase decreased (Investigations) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 4 | 1 | 0
Aspartate aminotransferase decreased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 1 | 0
Bilirubin conjugated increased (Investigations) | 1 | 0 | 1
Blood albumin decreased (Investigations) | 1 | 0 | 0
Blood alkaline phosphatase decreased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 1 | 1
Blood bilirubin unconjugated increased (Investigations) | 1 | 0 | 1
Blood calcium decreased (Investigations) | 1 | 0 | 0
Blood cholesterol increased (Investigations) | 1 | 0 | 0
Blood phosphorus decreased (Investigations) | 1 | 0 | 0
Blood potassium decreased (Investigations) | 2 | 0 | 0
Carcinoembryonic antigen increased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 6 | 1 | 1
Platelet count decreased (Investigations) | 2 | 0 | 0
Protein total decreased (Investigations) | 2 | 0 | 0
Protein urine present (Investigations) | 1 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 1 | 0 | 0
Staphylococcus test positive (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0
White blood cell count decreased (Investigations) | 6 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 8 | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cholinergic syndrome (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 2 | 1 | 0
Adenomyosis (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Based on available preliminary data from phase I clinical studies (1412.1 and 1412.3), the decision was made to stop BI 905711 (TRAILR2/CDH17) development program. This decision is not related to any safety concerns or unfavorable benefit/risk balance, but to the lack of predictive biomarkers and the limited efficacy particularly in the context of the evolving treatment landscape for advanced colorectal cancer (CRC) and other gastrointestinal (GI) cancers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/92/NCT05087992/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-05): https://cdn.clinicaltrials.gov/large-docs/92/NCT05087992/SAP_001.pdf